CLINICAL TRIAL: NCT03803865
Title: A Randomized Controlled Trial Comparing a 30 Day Mediation App to 30 Day Active Problem Solving App: Stress Management in Customer Service Representatives
Brief Title: 30 Day Mobile App Programs for Stress Management in Customer Service Representatives
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carnegie Mellon University (Other)
Collaborators: Headspace Meditation Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: FP00000925
Record Dates: First submitted 2018-11-13; First posted 2019-01-15 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Psychological Stress; Inflammation
Keywords: Job Stress; Mindfulness; Inflammation; Neuroimaging
MeSH Terms: conditions — Stress, Psychological; Inflammation; Occupational Stress

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor will remain masked to which program the participant will use. However the experimenter will be helping set up the participants with the app content and thus will not be masked to condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Headspace (Active Comparator): 30-day smartphone based mindfulness training intervention consisting of 10-minutes for the first 10 days, 15 minutes for the next 10 days, and 20 minutes for the final 10 days.
  Interventions: Behavioral: Mindfulness Training
- Recharge (Active Comparator): 30-day smartphone based reflection and problem solving training intervention consisting of 10-minutes for the first 10 days, 15 minutes for the next 10 days, and 20 minutes for the final 10 days.
  Interventions: Behavioral: Reflection and Problem Solving

INTERVENTIONS:
Behavioral: Mindfulness Training — Guided mindfulness meditation and stress management training
  Arms: Headspace
Behavioral: Reflection and Problem Solving — Guided reflection,problem solving,and analytical thinking training
  Arms: Recharge

SUMMARY:
Burnout and stress at work can make individuals less productive, which can carry over into their personal and at-home lives and negatively impact health. Customer service representatives are under especially high strain as they are exposed to significant interpersonal conflict at work, both with frustrated customers and with pressure from coworkers and supervisors. However, recent research has found that different stress management interventions (e.g., mindfulness meditation training) can increase job satisfaction and work productivity. However, individuals with significant stress might find these training program classes difficult to attend with their busy schedules. Newer interventions have focused on smartphone mobile applications as an effective delivery system for these training programs. Thus, the purpose of this project is to conduct a randomized controlled trial (RCT) comparing two different stress management smartphone app programs to evaluate effects on job-related outcomes, functional and structural brain outcomes, and biology.

DETAILED DESCRIPTION:
Approach: Employees will be given study flyers describing the study and encouraged to call a project hotline to evaluate their study eligibility. Eligible participants will be scheduled for an in-person study baseline and neuroimaging appointment at Carnegie Mellon University where they will provide written informed consent, complete baseline survey measures, provide several drops of blood via a finger prick (Dried Blood Spot (DBS) samples), and complete a 60-minute neuroimaging scan. After completing baseline measures participants will be instructed on how to download and use the Headspace smartphone app, and will be randomly assigned to one of the two programs. Participants will be asked to complete a 7- minute end-of-day daily diary measure each day during the treatment period, which will measure stress, affect, sleep, and workplace perceptions (a text message link will be sent an hour before the participant's standard bedtime each day). The project team will monitor treatment adherence (participants who do not complete a daily practice session will be called and reminded the following day). In the week following the end of the treatment period, participants will be scheduled to come back to Carnegie Mellon for a post-treatment appointment where they will complete the same measures as at baseline (survey measures, DBS, and neuroimaging). Participants will then be debriefed, compensated, and dismissed. Approximately two months after participants complete the 30-day program, we will call them for a 15-minute follow-up call. During this call, participants will answer a few questionnaire items and a brief program evaluation.

Interventions: Participants will be asked to complete one lesson daily for 30- days on the Headspace app; the first ten lessons will be 10 minutes long, the next ten will be 15 minutes long, and the final ten will be 20 minutes long. The mindfulness program will consist of the standard base program offered in Headspace. The Recharge program will consist of problem solving and stress management instruction.

Setting and Participants: David Creswell's Health and Human Performance Laboratory at Carnegie Mellon University will direct this study. Participants will be customer service employees (those who interact with customers daily via phone or in-person interactions) recruited from the Pittsburgh region.

ELIGIBILITY:
Inclusion Criteria:

Fluent in English

* 18-70 years old
* Planning to remain in the Pittsburgh area for the duration of participation
* Endorse significant work stress

Exclusion Criteria:

* Any significant mental and physical health conditions
* Metal implants
* Significant claustrophobia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-02-07 (Actual); Primary Completion 2019-11-04 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Burnout | Change in burnout over 30 day period and 90 day post-intervention follow-up
  Evaluated using a burnout scale for customer service representatives. This scale is used to measures feelings of burnout, a psychological disposition characterized by emotional exhaustion, lack of personal accomplishment, and a tendency to depersonalize others. The 24-item scale uses a 6-point Likert scale, and items are summed to create a composite score, with a range of 24-144, higher scores indicating greater burnout.
  Analyses will focus on a time (baseline, post-intervention, follow-up) by group interaction, and subsequent within group and within timepoint main effects. Here we hypothesize that while there will be a main effect of time, there will be a significant time by group interaction on reducing burnout.
Job Stress | Change in job stress over 30 day period and 90 day post-intervention follow-up
  Evaluated using Job Content Questionnaire. The Job Content Questionnaire is designed to measure the social and psychological characteristics of the workplace environment such as psychological demands, decision latitude, social support, physical demands, and job insecurity. The Job Stress measure will be calculated by combining the Psychological Demands and Decision Latitude subscales. The Psychological Demands subscale is 5-items and the Decision Latitude is 9-items. All are scored on a 1-4 Likert, resulting in a range of 14-56, scored such that higher numbers indicate greater job stress.
  Analyses will focus on a time (baseline, post-intervention, follow-up) by group interaction, and subsequent within group and within timepoint main effects. Here we hypothesize that while there will be a main effect of time, there will be a significant time by group interaction on reducing job stress.
Job Satisfaction | Change in job satisfaction over 30 day period.
  Evaluated using Job Satisfaction Questionnaire. This is a 10-item scale, each item scored on a 1-5 Likert scale, resulting in a range of 10-50, with higher scores indicating greater job satisfaction as follows:
  * 10-26: very low satisfaction
  * 27-31: low satisfaction
  * 32-38: average satisfaction
  * 39-41: high satisfaction
  * 42-50: very high satisfaction
  Analyses will focus on a time (baseline, post-intervention, follow-up) by group interaction, and subsequent within group and within timepoint main effects. Here we hypothesize that while there will be a main effect of time, there will be a significant time by group interaction on increasing job satisfaction.
Work Life Conflict | Change in work-life conflict over 30 day period.
  Evaluated using Work Life Conflict Scale.The Work Life Conflict designed to measure conflict between work and non-work experiences. The 5-item measure has been used in previous work, and participants respond to each item using a 1-7 Likert scale with higher numbers indicating greater work-life conflict. Some previous work has averaged responses to the 5-items, thus resulting in a range of 1-7 for this scale.
  Analyses will focus on a time by group interaction, and subsequent within group and within timepoint main effects. Here we hypothesize that while there will be a main effect of time, there will be a significant time by group interaction on reducing work-life conflict.
Life Work Conflict | Change in life-work conflict over 30 day period.
  Evaluated using Life Work Conflict Scales.The Life Work Conflict designed to measure conflict between non-work experiences and the individual's experiences at work. The 5-item measure has been used in previous work, and participants respond to each item using a 1-7 Likert scale with higher numbers indicating greater life-work conflict. Some previous work has averaged responses to the 5-items, thus resulting in a range of 1-7 for this scale.
  Analyses will focus on a time by group interaction, and subsequent within group and within timepoint main effects. Here we hypothesize that while there will be a main effect of time, there will be a significant time by group interaction on reducing life-work conflict.
Number of Sick Days taken | 2-month post-intervention follow-up
  Evaluated by asking at 2-month post-intervention follow-up.
  Analyses will focus on a main effect of group on lower number of sick days taken.
Functional neural activity to Positive Stimuli | Change in functional neural activity over 30 day period.
  Functional neural activity to a task displaying positive vs. neutral images. Analyses will focus on a time (baseline, post-intervention) by group (Headspace, Recharge) interaction, and subsequent within group and within timepoint main effects. ROI and connectivity analyses will focus on the reward network. Correlations with changes in included questionnaires and biology will also be assessed.
Functional neural activity to Negative Stimuli | Change in functional neural activity over 30 day period.
  Functional neural activity to a task displaying negative vs. neutral images. Analyses will focus on a time (baseline, post-intervention) by group (Headspace, Recharge) interaction, and subsequent within group and within timepoint main effects. ROI and connectivity analyses will focus on the threat/salience network. Correlations with changes in included questionnaires and biology will also be assessed.
Resting state functional connectivity | Change in resting state functional connectivity over 30 day period.
  Resting state functional connectivity will also be assessed using a time by group interaction and time and group main effects. We will conduct analyses focusing on the default mode and frontostriatal networks. Correlations with changes in included questionnaires and biology will also be assessed.
Diffusion Spectrum Imaging (DSI): Assess change in brain white matter tracts | Change in white matter integrity over 30 day period.
  Diffusion spectrum analyses will include time x group changes in white matter using fractional anisotropy (FA). Analyses will focus on whole brain FA (i.e., white matter integrity across the whole brain). Further analyses will explore associations between changes in white matter and our other outcomes of interest (behavior, biology, affect, functional task performance, etc.).
Changes in Amygdala Volume | Change in amygdala volume over 30 day period.
  Structural changes in the amygdala will also be assessed using time by group interaction and time and group main effects. Voxel based morphometry techniques will be used. In particular, change in gray matter volume will also be correlated with our relevant outcomes to assess whether changes in structure are associated with important changes in behavior, biology or affect.
Changes in Reward Network Volume | Change in brain volume over 30 day period.
  Structural changes in the reward network will also be assessed using time by group interaction and time and group main effects. Voxel based morphometry techniques will be used. In particular, these changes in gray matter volume will also be correlated with our relevant outcomes to assess whether changes in structure are associated with important changes in behavior, biology or affect.
Inflammatory Gene Expression | Change in gene expression over 30 day period.
  Changes in gene expression will be assessed using a time by group interaction (with time and group main effects also examined as ancillary findings, and in the event a significant time by group interaction is observed, follow-up group-stratified "simple effects" analyses of time effects may also be conducted to help interpret results). Analyses will focus an a priori-specified gene regulation pattern involving increased expression of inflammation-related genes and decreased expression of antiviral gene - a pattern called the conserved transcriptional response to adversity (CTRA).
Daily Diary--Change in self-reported productivity at work | Assessed daily to assess change in self-reported productivity during 30 day intervention
  Measures will be assessed end-of-day ("I was productive at work today." on 1-7 agreement Likert scale). Analyses will use multilevel modeling to explore differences between groups. Here, we will explore a possible time by group interaction on increased productivity.
Daily Diary--Change in self-reported engagement in meaningful activities at work | Assessed daily to assess change in engagement of meaningful activities during 30 day intervention
  Measures will be assessed end-of-day ("I feel like I did something meaningful at work today." on 1-7 agreement Likert scale). Analyses will use multilevel modeling to explore differences between groups. Here, we will explore a possible time by group interaction on increased self-reports of meaningful activities at work.
Daily Diary--Change in self-reported attention at work | Assessed daily to assess change in self-reported attention at work during 30 day intervention
  Measures will be assessed end-of-day ("At work today, I found myself doing things without really paying attention." adapted from Mindful Attention and Awareness Scale, answered on 1-6 frequency scale). Analyses will use multilevel modeling to explore differences between groups. Here, we will explore a possible time by group interaction on increased attention at work.
Daily Diary--Interpersonal conflict with customers and coworkers | Assessed daily to assess change in interpersonal conflict during 30 day intervention
  Interpersonal conflict with customers and coworkers will be assessed by the following questions (1-"none at all" to 5-"a great deal" scale):
  * How much conflict did you experience with customers today?
  * How much conflict with coworkers and managers/supervisors did you experience today?
  These items were selected to capture the listed outcome measure and do not come from a previously used scale. The outcome measure will be assessed end-of-day during the 30 day period.
  Analyses will use multilevel modeling to explore differences between groups. Here, we will explore a possible time by group interaction on reduced interpersonal conflict with customers and coworkers.
Daily Diary--Change in perceived stress at work | Assessed daily to assess change in perceived stress during 30 day intervention
  Measures will be assessed end-of-day using three items from Perceived Stress Scale adapted for work. Answered on a 0-never to 4-very often scale, with higher scores indicating greater perceived stress at work. Analyses will use multilevel modeling to explore differences between groups. We hypothesize a main effect of time, and a possible time by group interaction effect on perceived stress.

SECONDARY OUTCOMES:
Perceived Stress | Change in perceived stress over 30 day period.
  Evaluated using Perceived Stress Scale (PSS). The PSS measures the degree to which situations in one's life are appraised as stressful. Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress.
  * Scores ranging from 0-13 would be considered low stress.
  * Scores ranging from 14-26 would be considered moderate stress.
  * Scores ranging from 27-40 would be considered high perceived stress.
  Here, we expect a main effect of time, with a possible time by group interaction on lowered perceived stress.
Self-reported physical health | Change in self-reported physical over 30 day period.
  Evaluated using the SF-12, a 12-item scale assessing physical health and mental health. Composite scores range from 0-100 with higher scores indicating better health.
  Here, we expect a main effect of time, with a possible time by group interaction on improved self-reported physical health.
Self-reported depressive symptoms | Change in self-reported depressive symptoms over 30 day period.
  Evaluated using the CES-D which measures depressive symptoms over the last two weeks using 20-items. The total score is a sum of the items and scores can range from 0-60, with higher scores indicating greater depressive symptoms. A score equal to or above 16 can indicate a person at risk for clinical depression.
  Here, we expect a main effect of time, with a possible time by group interaction on lowered depressive symptoms
Mindfulness | Change in mindfulness over 30 day period.
  Evaluated using the Five Factor Mindfulness Questionnaire (FFMQ). This FFMQ is based on a factor analytic study of five independently developed mindfulness questionnaires. The analysis yielded five factors that appear to represent elements of mindfulness as it is currently conceptualized. The five facets are observing, describing, acting with awareness, non-judging of inner experience, and non-reactivity to inner experience. The 39-item scale is scored on 1-very rarely true to 5-very often true scale, range 39-195, with higher scores indicating greater mindfulness.
  Here, we expect a time by group interaction on increased mindfulness.
Social Support Perceptions | Change in social support perceptions over 30 day period.
  Evaluated using the Social Provisions Scale.The Social Provisions Scale was developed to assess the provisions of social relationships and what we receive from relationships with other people. The six provisions include guidance (advice or information), reliable alliance (assurance that others can be counted on in times of stress), reassurance of worth (recognition of one's competence), attachment (emotional closeness), social integration (a sense of belonging to a group of friends), and opportunity for nurturance (providing assistance to others) across 24 items. These subscales are summed to create a score for each subscale (range of 4-16), and subscales are summed together to create a composite total score (range of 24-96) with higher scores indicating higher perceptions of social support.
  Here, we will explore a possible time by group interaction on increased perceptions of available social support.
Loneliness | Change in self-reported loneliness over 30 day period.
  Evaluated using the UCLA Loneliness Scale. The UCLA Loneliness scale is designed to measure one's subjective feelings of loneliness as well as feelings of social isolation. Scores are summed from each item and higher scores indicate greater degrees of loneliness (range 20-80).
  Here, we will explore a possible time by group interaction on reduced loneliness.
Distress Tolerance/Acceptance | Change distress tolerance/acceptance over 30 day period.
  Evaluated using the Distress Tolerance Scale which assesses the perceived ability to tolerate distress using 16-items, summed, with a range of 16-90 with higher scores indicating greater levels of distress tolerance.
  Here, we will explore a possible time by group interaction on increased acceptance.
Equanimity | Change in equanimity over 30 day period.
  Evaluated using the White Bear Thought Suppression Inventory. 15 items answered on a 5-point Likert scale and summed, resulting in a range of 15-75 (higher scores indicating greater thought suppression). Greater thought suppression is believed to be an indicator of low equanimity.
  Here, we will explore a possible time by group interaction on increased equanimity (reduced thought suppression scores).
C-reactive protein (CRP) levels | Change in C-Reactive Protein levels over 30 day period.
  CRP levels will be assessed through dried blood spots collected at baseline and post-intervention. Changes in CRP levels will be assessed using a time by group interaction and time and group main effects. We hypothesize a main effect of time, with exploratory analyses to examine the interaction effect.

OTHER OUTCOMES:
Daily Diary--Positive Affect | Assessed daily during 30 day intervention
  Measures will be assessed end-of-day ("How positive was your mood today?" on 1-not at all to 7-extremely scale). Analyses will use multilevel modeling to explore differences between groups. We hypothesize a time by group interaction effect on positive affect.
Daily Diary--Negative Affect | Assessed daily during 30 day intervention
  Measures will be assessed end-of-day ("How positive was your mood today?" on 1-not at all to 7-extremely scale). Analyses will use multilevel modeling to explore differences between groups. We hypothesize a main effect of time on negative affect.
Daily Diary--Self-reported feelings about work shift | Assessed daily during 30 day intervention
  Measures will be assessed end-of-day ("Rate how you feel about today's shift at work." on a 1-extremely bad to 7-extremely good scale). Analyses will use multilevel modeling to explore differences between groups. Here, we will explore a possible time by group interaction on more positive feelings about work.
Daily Diary--Self-reported positive attitude at work | Assessed daily during 30 day intervention
  Measures will be assessed end-of-day ("I had a positive attitude at work today." on a 1-7 agreement Likert scale). Analyses will use multilevel modeling to explore differences between groups. Here, we will explore a possible time by group interaction on increased positive attitude at work.
Daily Diary--Feelings of acceptance at work | Assessed daily during 30 day intervention
  Measures will be assessed end-of-day using one item from the Philadelphia Mindfulness Scale ("There were things I tried not to think about while I was at work today." reverse scored such that higher scores reflect more acceptance). Analyses will use multilevel modeling to explore differences between groups. Here, we will explore a possible time by group interaction on increased acceptance.
Daily Diary- Work-life conflict | Assessed end-of-day during 30 day intervention
  Measures will be assessed end-of-day ("The demands of my work interfered with my life away from work today." on a 1-7 agreement Likert scale). Analyses will use multilevel modeling to explore differences between groups. Here, we will explore a possible time by group interaction on reduced work-life conflict.
Daily Diary- Life-Work conflict | Assessed daily during 30 day intervention
  Measures will be assessed end-of-day ("Personal life issues interfered with my ability to perform work-related duties today." on a 1-7 agreement Likert scale). Analyses will use multilevel modeling to explore differences between groups. Here, we will explore a possible time by group interaction on reduced life-work conflict.
Daily Diary- Number of social interactions at work and outside of work | Assessed daily during 30 day intervention
  Measures will be assessed end-of-day. Analyses will use multilevel modeling to explore differences between groups. Here, we will explore a possible time by group interaction on a higher number of social interactions outside of work.
Daily Diary--Social Connection | Assessed end-of-day during 30 day intervention
  Measures will be assessed end-of-day and ask the participant to reflect on how connected they felt that day. Analyses will use multilevel modeling to explore differences between groups. Here, we will explore a possible time by group interaction on increased feelings of social connection.
Daily Diary--Self-reported number of hours of sleep | Assessed daily during 30 day intervention
  Measures will be assessed end-of-day. Analyses will use multilevel modeling to explore differences between groups. We hypothesize a main effect of time, and a possible time by group interaction effect on increased hours asleep.

CONTACTS AND LOCATIONS:
Overall Officials: David Creswell, Ph.D, Study Chair — Carnegie Mellon University
Locations (1):
- Carnegie Mellon University, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The research team will share data associated with self-reports (e.g. job satisfaction, stress levels) and gene expression assays. All data and documentation will be de-identified and will be consistent with applicable laws and regulations. Neuroimaging data will be defaced such that no identifiable information remains on the images.When publishers require analyzed data to be available in order to publish manuscripts, those data will be provided by link to the repository. Data will be shared via KiltHub, a comprehensive repository hosted by Carnegie Mellon University. Data will be shared when a publisher requests that information be shared as part of the terms of publication. A file containing all variables necessary to replicate the analyses from the manuscript will be uploaded. If neuroimaging data is to be shared, the relevant scan will be shared after being de-identified, in addition to the necessary structural scan (as it is required for preprocessing co-registration).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Study data will become available when journals ask for these items upon publication of a paper from this dataset.
Access Criteria: Data relevant to replicating analyses will be shared via KiltHub, a comprehensive repository hosted by Carnegie Mellon University. This repository helps keep track of who has accessed data, and is supported by the university and thus be available to other researchers.

REFERENCES:
- [Background] Slutsky J, Chin B, Raye J, Creswell JD. Mindfulness training improves employee well-being: A randomized controlled trial. J Occup Health Psychol. 2019 Feb;24(1):139-149. doi: 10.1037/ocp0000132. Epub 2018 Oct 18. PMID 30335419
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Russell D, Peplau LA, Cutrona CE. The revised UCLA Loneliness Scale: concurrent and discriminant validity evidence. J Pers Soc Psychol. 1980 Sep;39(3):472-80. doi: 10.1037//0022-3514.39.3.472. PMID 7431205
- [Background] Wegner DM, Zanakos S. Chronic thought suppression. J Pers. 1994 Dec;62(4):616-40. doi: 10.1111/j.1467-6494.1994.tb00311.x. PMID 7861307
- [Background] Singh, J., Goolsby, J. R., & Rhoads, G. K. (1994). Behavioral and psychological consequences of boundary spanning burnout for customer service representatives. Journal of Marketing Research, 558-569.
- [Background] Schnall PL, Schwartz JE, Landsbergis PA, Warren K, Pickering TG. A longitudinal study of job strain and ambulatory blood pressure: results from a three-year follow-up. Psychosom Med. 1998 Nov-Dec;60(6):697-706. doi: 10.1097/00006842-199811000-00007. PMID 9847028
- [Background] Macdonald, S., & Maclntyre, P. (1997). The generic job satisfaction scale: Scale development and its correlates. Employee Assistance Quarterly, 13(2), 1-16.
- [Background] Waumsley, J. A., Houston, D. M., & Marks, G. (2010). What about us? Measuring the work- life balance of people who do not have children. Review of European Studies , 2(2), 3- 17.
- [Background] Cole SW, Conti G, Arevalo JM, Ruggiero AM, Heckman JJ, Suomi SJ. Transcriptional modulation of the developing immune system by early life social adversity. Proc Natl Acad Sci U S A. 2012 Dec 11;109(50):20578-83. doi: 10.1073/pnas.1218253109. Epub 2012 Nov 26. PMID 23184974
- [Background] Brown KW, Ryan RM. The benefits of being present: mindfulness and its role in psychological well-being. J Pers Soc Psychol. 2003 Apr;84(4):822-48. doi: 10.1037/0022-3514.84.4.822. PMID 12703651
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Background] Radloff, L.S. The CES-D Scale: A self-report depression scale for research in the general population. Applied Psychological Measurement, 1977.
- [Background] Baer RA, Smith GT, Hopkins J, Krietemeyer J, Toney L. Using self-report assessment methods to explore facets of mindfulness. Assessment. 2006 Mar;13(1):27-45. doi: 10.1177/1073191105283504. PMID 16443717
- [Background] Cutrona, C. E., & Russell, D. W. (1987). The provisions of social relationships and adaptation to stress. Advances in personal relationships, 1(1), 37-67.
- [Background] Simons, J. S., & Gaher, R. M. (2005). The Distress Tolerance Scale: Development and validation of a self-report measure. Motivation and Emotion, 29(2), 83-102.
- [Background] Cardaciotto L, Herbert JD, Forman EM, Moitra E, Farrow V. The assessment of present-moment awareness and acceptance: the Philadelphia Mindfulness Scale. Assessment. 2008 Jun;15(2):204-23. doi: 10.1177/1073191107311467. Epub 2008 Jan 9. PMID 18187399